CLINICAL TRIAL: NCT06060262
Title: The Clinical Significance of Metabolic Adipo-myokines and Alterations of Body Composition in Patients With End Stage Lung Cancer
Brief Title: The Alterations of Metabolic Adipo-myokines and Body Composition in End Stage Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202201448B0
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer Metastatic
Keywords: adipo-myokines; body composition; end stage lung cancer; clinical outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Adipo-myokines concentrations will be checked using residual plasma specimens on the date of before therapy, 4 weeks after therapy and 12 weeks after therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators conduct this prospective study and wish to elucidate the association of serial change of body composition, serum adipo-myokines and adverse effect of chemotherapy and lung cancer prognosis

DETAILED DESCRIPTION:
Recently, the skeletal muscle was viewed as having biochemical function in additional to traditional biomechanical function. What's more important is that muscles could synthesize and release adipo-myokines during contraction. The adipo-myokines can affect muscle regeneration, muscle atrophy, muscle mass, autophagy, fatty acid oxidation and mitochondrial biosynthesis.Studies have also found that exercise can promote the function of macrophages and regulate both pro-inflammatory and anti-inflammatory phenotypes, helping the body to establish a stable immune balance.

Since body composition can illustrate malnutrition status and cancer cachexia present, and body composition can be affected by serum adipo-myokines level. Therefore, the investigators conduct this study and wish to see the association of serial body composition and serum adipo-myokines changes with lung cancer clinical outcomes and adverse effect of any anti-cancer regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of lung cancer stage III to stage IV
2. Adults over 20 years old
3. Daily performance status of 0- 2

Exclusion Criteria:

1. Cardiac stents or pacemakers

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who diagnosed with lung cancer including small cell and non-small cell lung cancer from 2023-03-1to 2026-02-28 will be eligible for the study. Every patients' performance status must be in 0-2 and can receive any cancer treatments including chemotherapy.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of white blood cell change among before, during and after cancer therapy | week 0 , week 4 and week 12 after cancer theraphy
  assessing the change of white blood cell count among week 0, week 4 and week 12
Percentage of body fat change among before, during and after cancer therapy | week 0 , week 4 and week 12 after cancer theraphy
  assessing the change of percentage of body fat among week 0, week 4 and week 12
Percentage of total body water change among before, during and after cancer therapy | week 0 , week 4 and week 12 after cancer theraphy
  assessing the change of total body water percentage among week 0, week 4 and week 12
Percentage of soft lean mass change among before, during and after cancer therapy | week 0 , week 4 and week 12 after cancer theraphy
  assessing the change of soft lean mass percentage among week 0, week 4 and week 12
Concentration of plasma CEA change among before, during and after cancer therapy | week 0, week 4 and week 12 after cancer theraphy
  assessing the change of plasma CEA concentration among week 0, week 4 and week 12
Concentration of plasma albumin change among before, during and after cancer therapy | week 0 , week 4 and week 12 after cancer theraphy
  assessing the change of plasma albumin concentration among week 0, week 4 and week 12
Concentration of plasma myostatin change among before, during and after cancer therapy | week 0 , week 4 and week 12 after cancer theraphy
  assessing the change of plasma myostatin concentration among week 0, week 4 and week 12
Concentration of plasma FSTL-1 change among before, during and after cancer therapy | week 0 , week 4 and week 12 after cancer theraphy
  assessing the change of plasma FSTL-1 concentration among week 0, week 4 and week 12
Concentration of plasma IL-6 change among before, during and aftercancer therapy | week 0 , week 4 and week 12 after cancer theraphy
  assessing the change of plasma IL-6 concentration among week 0, week 4 and week 12
Concentration of plasma irisin change among before, during and after cancer therapy | week 0 , week 4 and week 12 after cancer theraphy
  assessing the change of plasma irisin concentration among week 0, week 4 and week 12
Concentration of plasma adiponectin change among before, during and after cancer therapy | week 0 , week 4 and week 12 after cancer theraphy
  assessing the change of plasma adiponectin concentration among week 0, week 4 and week 12
Concentration of plasma MCP-1 change among before, during and after cancer therapy | week 0 , week 4 and week 12 after cancer theraphy
  assessing the change of plasma MCP-1 concentration among week 0, week 4 and week 12
Concentration of plasma aquaporin change among before, during and after cancer therapy | week 0 , week 4 and week 12 after cancer theraphy
  assessing the change of plasma aquaporin concentration among week 0, week 4 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: TSENG CHIA-CHENG, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No